CLINICAL TRIAL: NCT01334918
Title: A Phase 2, Open-Label, Randomized, Cross-Over Study of Regadenoson in Subjects Undergoing Stress Myocardial Perfusion Imaging by Multidetector Computed Tomography (MDCT) and Single Photon Emission Computed Tomography (SPECT)
Brief Title: A Study of Regadenoson in Subjects Undergoing Stress Myocardial Perfusion Imaging (MPI) Using Multidetector Computed Tomography (MDCT) Compared to Single Photon Emission Computed Tomography (SPECT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 3606-CL-2001
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: pharmacologic stress; Coronary Artery Disease (CAD); regadenoson; ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia | interventions — regadenoson; Technetium Tc 99m Sestamibi; technetium tc-99m tetrofosmin; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Photon Emission Computed Tomography (SPECT) (Experimental): Resting SPECT imaging was performed prior to regadenoson stress SPECT
  imaging. Imaging was conducted with one of two radiotracers (99mTc sestamibi or tetrofosmin). Regadenoson 0.4 mg was administered prior to stress SPECT as a single bolus injection.
  Interventions: Drug: regadenoson; Radiation: technetium Tc99m sestamibi /technetium Tc99m tetrafosmin; Radiation: Contrast; Procedure: Single Photon Emission Computed Tomography; Procedure: Multidetector Computed Tomography
- Multidetector Computed Tomography (MDCT) (Experimental): Multidetector Computed Tomography (MDCT), composed of CCTA and regadenoson CTP. Regadenoson stress CTP was performed prior to rest CCTA/CTP imaging. Regadenoson 0.4 mg was administered prior to stress CTP as a single bolus injection. The rest CCTA/CTP was performed at least 30 minutes after completion of the stress CTP, after resolution of any symptoms brought on by the regadenoson infusion and after the participant's heart rate had returned to baseline.
  Interventions: Drug: regadenoson; Radiation: technetium Tc99m sestamibi /technetium Tc99m tetrafosmin; Radiation: Contrast; Procedure: Single Photon Emission Computed Tomography; Procedure: Multidetector Computed Tomography

INTERVENTIONS:
Drug: regadenoson — Administered by intravenous bolus.
  Other Names: CVT 3146; Lexiscan
Radiation: technetium Tc99m sestamibi /technetium Tc99m tetrafosmin — Administered by intravenous infusion
  Other Names: Cardiolite; Myoview
Radiation: Contrast — Administered by intravenous infusion.
Procedure: Single Photon Emission Computed Tomography — Procedure/Surgery
Procedure: Multidetector Computed Tomography — Procedure/Surgery

SUMMARY:
The purpose of this study is to compare Multidetector Computed Tomography (MDCT) and Single Photon Emission Computed Tomography (SPECT) stress myocardial perfusion imaging (MPI) with regadenoson in order to detect the presence or absence of reversible defects.

DETAILED DESCRIPTION:
All participants will be randomized to one of two imaging sequences: rest/stress SPECT on Day 1 followed by stress/rest MDCT on Day 2 or stress/rest MDCT on Day 1 followed by rest/stress SPECT on Day 2. All stress scans will involve the injection of regadenoson as the pharmacologic stress agent.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects must be ≥ 45 years of age
* Female subjects must be ≥ 50 years of age
* Subject has met at least one of the following three criteria:

  * has a suspected (clinical impression) or known diagnosis of coronary artery disease (CAD) with typical angina that has been referred from nuclear cardiology lab schedule or cardiac computed tomography (CT) schedule
  * has stable symptoms with possible elective catheterization procedure scheduled and where further imaging may be beneficial;
  * has known CAD from a previous invasive coronary angiography (ICA) performed more than 12 weeks prior to screening who now present with new cardiac symptoms
* Subject has been referred for a clinically indicated myocardial perfusion imaging procedure or Cardiac CT procedure for suspected moderate or high risk CAD
* Subject must abstain from eating and drinking 30 minutes prior and 30 minutes post study drug administration
* Subject must abstain from smoking 3 hours prior and 8 hours post study drug administration
* Subject must abstain from any intake of methylxanthine-containing foods and beverages within 12 hours prior to Day 1 visit through the Day 3 Follow-Up Visit, as these foods may alter regadenoson effects. Subject is able to safely abstain from theophylline use for 12 hours prior to study drug administration

Exclusion Criteria:

* Subject is concurrently participating in another drug study or has received an investigational drug within 30 days prior to Screening
* Subject has a history of a clinically significant illness (other than CAD), medical condition, or laboratory abnormality, which would preclude participation in the study
* Subject has renal dysfunction demonstrated by a glomerular filtration rate (GFR) < 45 mL/min (calculated using Cockroft-Gault formula Note: Subjects with a GFR 45-60 mL/min will undergo a hydration procedure
* Female subject who is pregnant, lactating or of childbearing potential that refuses to use a medically acceptable form of contraception until the Telephone Follow up Visit is complete
* Female subject has a positive pregnancy test prior to randomization
* Subject has a history of second or third degree heart block or sinus node dysfunction unless the subject has a functioning pacemaker
* Subject has symptomatic hypotension (temporary and reversible conditions that no longer exist are allowed)
* Subject is allergic or intolerant to aminophylline, nitroglycerin or metoprolol
* Subject is allergic or intolerant to regadenoson or any of its excipients
* Subject is unable or unwilling to comply with the procedure schedule
* Subject has previously enrolled in this study or was enrolled in another regadenoson study sponsored by Astellas
* Subject has atrial fibrillation or significant arrhythmias which may result in decreased image quality for the imaging studies (CT and SPECT)
* Subject has high heart rate (> 65 beats per minute) and contra-indications to administer beta-blockers (severe chronic obstructive pulmonary disease (COPD) or asthma, second and third degree atrioventricular block)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-04-26 (Actual); Primary Completion 2012-07-02 (Actual); Study Completion 2012-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (11):
- United States (11):
  - Sutter Roseville Medical Center, Roseville, California
  - Harbor UCLA Medical Center, Torrance, California
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Midwest Cardiology Associates, P.C., Overland Park, Kansas
  - Maine Research Associates, Auburn, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Cury RC, Kitt TM, Feaheny K, Akin J, George RT. Regadenoson-stress myocardial CT perfusion and single-photon emission CT: rationale, design, and acquisition methods of a prospective, multicenter, multivendor comparison. J Cardiovasc Comput Tomogr. 2014 Jan-Feb;8(1):2-12. doi: 10.1016/j.jcct.2013.09.004. Epub 2013 Oct 18. PMID 24314823
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=225

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: SPECT - MDCT: Day 1: a rest Single Photon Emission Computed Tomography (SPECT) and a regadenoson stress SPECT procedure. Day 2: a regadenoson stress Computed Tomography Perfusion (CTP) and a rest Coronary Computed Tomography Angiography (CCTA)/CTP procedure. Regadenoson 0.4 mg was administered prior to each stress procedure as a single bolus injection.
- Sequence 2: MDCT - SPECT: Day 1: a regadenoson stress CTP and a rest CCTA/CTP procedure. Day 2: a rest SPECT and a regadenoson stress SPECT procedure. Regadenoson 0.4 mg was administered prior to each stress procedure as a single bolus injection.
Period: Overall Study
Arm/Group | Sequence 1: SPECT - MDCT | Sequence 2: MDCT - SPECT
Started | 63 | 61
Randomized + 1 Stress Scan | 57 (Equates to Safety Analysis Set (SAF)) | 61 (Equates to Safety Analysis Set (SAF))
Completed | 55 | 60
Not Completed | 8 | 1
Not completed — Did not receive study drug | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): All randomized participants who received at least 1 dose of regadenoson.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: SPECT - MDCT | Sequence 2: MDCT - SPECT | Total
Number analyzed (Participants) | 57 | 61 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.19) | 62.3 (9.41) | 61.6 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 39 | 46 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  White | 52 | 54 | 106
  Black or African American | 2 | 5 | 7
  Asian | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 37 | 41 | 78
  Hispanic or Latino | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reversible Defects
Description: The number of reversible defects categorized into absence or presence of ischemia (0-1 versus ≥2), as assessed by the central imaging laboratory for both SPECT and MDCT. The 17-segment model for standardized myocardial segmentation was used for myocardial perfusion readings for SPECT and MDCT. At rest and stress, each segment was scored on a 0 to 4 scale according to the amount of contrast or radiotracer the myocardium in the segment absorbed: -0: normal perfusion -1: slightly reduced contrast/radiotracer uptake -2: moderately reduced contrast/radiotracer uptake -3: severely reduced contrast/radiotracer uptake -4: absent contrast/radiotracer uptake. The median score from the 3 blinded readers for each segment was used. If the stress score was ≥ 2 and the rest score was less than the stress score, the segment was counted as having a reversible defect. A participant was classified as ischemic in the presence of 2 or more segments with reversible defects, excluding segment 17.
Time Frame: Day 1 and Day 2
Population: The number of participants analyzed represents the full analysis set, defined as all randomized patients with interpretable SPECT and CTP scans as determined by at least two of the three blinded readers.
Measure: Number; unit: participants
Groups:
- CTP: 0 - 1 Reversible Defects: Participants with 0 - 1 reversible defects as assessed by regadenoson stress computed tomography perfusion (CTP).
- CTP: ≥ 2 Reversible Defects: Participants with ≥ 2 reversible defects as assessed by regadenoson stress computed tomography perfusion (CTP).
- CTP: All Reversible Defects: All participants as assessed by regadenoson stress computed tomography perfusion (CTP).
Arm/Group | CTP: 0 - 1 Reversible Defects | CTP: ≥ 2 Reversible Defects | CTP: All Reversible Defects
Number analyzed (Participants) | 85 | 25 | 110
participants
  SPECT: 0-1 Reversible defects | 84 | 16 | 100
  SPECT: ≥ 2 Reversible defects | 1 | 9 | 10
  SPECT: All Reversible defects | 85 | 25 | 110
Statistical Analysis 1: Comparison: CTP: 0 - 1 Reversible Defects vs CTP: ≥ 2 Reversible Defects vs CTP: All Reversible Defects; Analysis of agreement rate based on participants with 0 -1 and ≥ 2 reversible defects according to SPECT. Agreement is defined as the proportion of participants who had the same status from SPECT and MDCT, averaged across those with 2 or more reversible defects and those without, where SPECT is the reference standard; Test type: Non-Inferiority or Equivalence — Predefined noninferiority criterion: If the lower boundary of the 95% CI was within 0.15 of 0.78, MDCT would be determined to be noninferior to SPECT; Agreement rate = 0.87, 95% CI 2-sided [0.77 to 0.97], Standard Error of Mean 0.051

2. Secondary Outcome: Overall Image Quality of Scans by Modality and Reviewer
Description: Overall image quality was assessed by three independent blinded readers for each modality (single photon emission computed tomography (SPECT) and multidetector computed tomography (MDCT)). Image quality was rated on a 4-point scale as either excellent, good, fair or poor at rest using SPECT and MDCT and under stress using regadenoson SPECT and regadenoson stress computed tomography perfusion (CTP).
Time Frame: Day 1 and Day 2
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: participants
Groups:
- SPECT: Reviewer 1: Analysis of image quality of single photon emission computed tomography (SPECT) images performed by SPECT Reviewer 1.
- SPECT: Reviewer 2: Analysis of image quality of single photon emission computed tomography (SPECT) images performed by SPECT Reviewer 2.
- SPECT: Reviewer 3: Analysis of image quality of single photon emission computed tomography (SPECT) images performed by SPECT Reviewer 3.
- MDCT: Reviewer 1: Analysis of image quality of multidetector computed tomography (MDCT) images performed by MDCT Reviewer 1.
- MDCT: Reviewer 2: Analysis of image quality of multidetector computed tomography (MDCT) images performed by MDCT Reviewer 2.
- MDCT: Reviewer 3: Analysis of image quality of multidetector computed tomography (MDCT) images performed by MDCT Reviewer 3.
Arm/Group | SPECT: Reviewer 1 | SPECT: Reviewer 2 | SPECT: Reviewer 3 | MDCT: Reviewer 1 | MDCT: Reviewer 2 | MDCT: Reviewer 3
Number analyzed (Participants) | 110 | 110 | 110 | 110 | 110 | 110
participants
  Rest: Excellent | 89 | 25 | 83 | 30 | 40 | 56
  Rest: Good | 16 | 53 | 23 | 56 | 37 | 43
  Rest: Fair | 4 | 31 | 4 | 23 | 33 | 11
  Rest: Poor | 1 | 1 | 0 | 1 | 0 | 0
  Stress: Excellent | 89 | 35 | 78 | 5 | 15 | 37
  Stress: Good | 16 | 51 | 27 | 48 | 24 | 36
  Stress: Fair | 4 | 24 | 5 | 56 | 62 | 34
  Stress: Poor | 1 | 0 | 0 | 1 | 9 | 3

3. Secondary Outcome: Number of Participants With Reversible Defects in the Left Anterior Descending Coronary Artery (LAD)
Description: The number of reversible defects in the LAD categorized into absence or presence of ischemia (0-1 versus ≥2), as assessed by the central imaging laboratory for both SPECT and MDCT. The 17-segment model for standardized myocardial segmentation was used for myocardial perfusion readings for SPECT and MDCT. At rest and stress, each segment was scored on a 0 to 4 scale according to the amount of contrast or radiotracer the myocardium in the segment absorbed: -0: normal perfusion -1: slightly reduced contrast/radiotracer uptake -2: moderately reduced contrast/radiotracer uptake -3: severely reduced contrast/radiotracer uptake -4: absent contrast/radiotracer uptake. The median score from 3 blinded readers for each segment was used. If the stress score was ≥ 2 and the rest score was less than the stress score, the segment was counted as having a reversible defect. A participant was classified as ischemic in the presence of ≥ 2 segments with reversible defects, excluding segment 17.
Time Frame: Day 1 and Day 2
Population: The number of participants analyzed represents the full analysis set where scans were available.
Measure: Number; unit: participants
Arm/Group | CTP: 0 - 1 Reversible Defects | CTP: ≥ 2 Reversible Defects | CTP: All Reversible Defects
Number analyzed (Participants) | 90 | 15 | 105
participants
  SPECT: 0 - 1 Reversible defects | 90 | 11 | 101
  SPECT: ≥ 2 Reversible defects | 0 | 4 | 4
  SPECT: All Reversible defects | 90 | 15 | 105

4. Secondary Outcome: Number of Participants With Reversible Defects in the Right Coronary Artery (RCA)
Description: The number of reversible defects in the RCA categorized into absence or presence of ischemia (0-1 versus ≥2), as assessed by the central imaging laboratory for both SPECT and MDCT. The 17-segment model for standardized myocardial segmentation was used for myocardial perfusion readings for SPECT and MDCT. At rest and stress, each segment was scored on a 0 to 4 scale according to the amount of contrast or radiotracer the myocardium in the segment absorbed: -0: normal perfusion -1: slightly reduced contrast/radiotracer uptake -2: moderately reduced contrast/radiotracer uptake -3: severely reduced contrast/radiotracer uptake -4: absent contrast/radiotracer uptake. The median score from 3 blinded readers for each segment was used. If the stress score was ≥ 2 and the rest score was less than the stress score, the segment was counted as having a reversible defect. A participant was classified as ischemic in the presence of ≥ 2 segments with reversible defects, excluding segment 17.
Time Frame: Day 1 and Day 2
Population: The number of participants analyzed represents the full analysis set where scans were available.
Measure: Number; unit: participants
Arm/Group | CTP: 0 - 1 Reversible Defects | CTP: ≥ 2 Reversible Defects | CTP: All Reversible Defects
Number analyzed (Participants) | 93 | 5 | 98
participants
  SPECT: 0 - 1 Reversible defects | 92 | 5 | 97
  SPECT: ≥ 2 Reversible defects | 1 | 0 | 1
  SPECT: All Reversible defects | 93 | 5 | 98

5. Secondary Outcome: Number of Participants With Reversible Defects in the Left Circumflex Coronary Artery (LCX)
Description: The number of reversible defects in the LCX categorized into absence or presence of ischemia (0-1 versus ≥2), as assessed by the central imaging laboratory for both SPECT and MDCT. The 17-segment model for standardized myocardial segmentation was used for myocardial perfusion readings for SPECT and MDCT. At rest and stress, each segment was scored on a 0 to 4 scale according to the amount of contrast or radiotracer the myocardium in the segment absorbed: -0: normal perfusion -1: slightly reduced contrast/radiotracer uptake -2: moderately reduced contrast/radiotracer uptake -3: severely reduced contrast/radiotracer uptake -4: absent contrast/radiotracer uptake. The median score from 3 blinded readers for each segment was used. If the stress score was ≥ 2 and the rest score was less than the stress score, the segment was counted as having a reversible defect. A participant was classified as ischemic in the presence of ≥ 2 segments with reversible defects, excluding segment 17.
Time Frame: Day 1 and Day 2
Population: The number of participants analyzed represents the full analysis set where scans were available.
Measure: Number; unit: participants
Arm/Group | CTP: 0 - 1 Reversible Defects | CTP: ≥ 2 Reversible Defects | CTP: All Reversible Defects
Number analyzed (Participants) | 92 | 13 | 105
participants
  SPECT: 0 - 1 Reversible defects | 90 | 9 | 99
  SPECT: ≥ 2 Reversible defects | 2 | 4 | 6
  SPECT: All Reversible defects | 92 | 13 | 105

6. Secondary Outcome: Number of Participants With Fixed Defects
Description: Using the 17-segment scoring system, a segment scored above 1 (i.e., 2 to 4) and equal at rest and stress was counted as having a fixed defect. At rest and stress, each segment was scored on a 0 to 4 scale according to the amount of contrast or radiotracer the myocardium in the segment absorbed: -0: normal perfusion -1: slightly reduced contrast/radiotracer uptake -2: moderately reduced contrast/radiotracer uptake -3: severely reduced contrast/radiotracer uptake -4: absent contrast/radiotracer uptake.
Time Frame: Day 1 and Day 2
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: participants
Groups:
- CTP: 0 Fixed Defects: Participants with zero fixed defects as assessed by regadenoson stress computed tomography perfusion (CTP).
- CTP: ≥ 1 Fixed Defects: Participants with ≥ 1 fixed defects as assessed by regadenoson stress computed tomography perfusion (CTP).
- CTP: All Fixed Defects: All participants as assessed by regadenoson stress computed tomography perfusion (CTP).
Arm/Group | CTP: 0 Fixed Defects | CTP: ≥ 1 Fixed Defects | CTP: All Fixed Defects
Number analyzed (Participants) | 95 | 15 | 110
participants
  SPECT: 0 Fixed Defects | 92 | 5 | 97
  SPECT: ≥ 1 Fixed Defects | 3 | 10 | 13
  SPECT: All Fixed Defects | 95 | 15 | 110
Statistical Analysis 1: Comparison: CTP: 0 Fixed Defects vs CTP: ≥ 1 Fixed Defects vs CTP: All Fixed Defects; Analysis of specificity based on participants with no fixed defects according to SPECT. Specificity is defined as a proportion of true negatives that are correctly identified, using SPECT as the reference standard; Test type: Superiority or Other; Specificity = 0.95, 95% CI 2-sided [0.90 to 0.99], Standard Error of Mean 0.022
Statistical Analysis 2: Comparison: CTP: 0 Fixed Defects vs CTP: ≥ 1 Fixed Defects vs CTP: All Fixed Defects; Analysis of sensitivity based on participants with ≥ 1 fixed defect according to SPECT. Sensitivity is the proportion of true positives that are correctly identified using SPECT as the reference standard; Test type: Superiority or Other; Sensitivity = 0.77, 95% CI 2-sided [0.54 to 1.00], Standard Error of Mean 0.117

7. Secondary Outcome: Percentage of Participants With Two or More Ischemic Segments on SPECT, But Less on CT
Description: Using SPECT as the reference standard, the false negative percentage was calculated as the percentage of participants with two or more ischemic segments on SPECT, but less on CT.
Time Frame: Day 1 and Day 2
Population: Full analysis set participants with two or more reversible defects.
Measure: Number; unit: percentage of participants
Groups:
- SPECT + MDCT: Participants underwent both a rest and stress SPECT series and a rest and stress MDCT series.
Arm/Group | SPECT + MDCT
Number analyzed (Participants) | 10
percentage of participants | 10

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were defined as adverse events observed from the time of administration of regadenoson to 24 hours after last study drug administration within each modality, i.e. from Day 1 to Day 3.
Description: Safety Analysis Set composed of all randomized patients who received at least 1 dose of regadenoson.
Groups:
- SPECT: Resting SPECT imaging was performed prior to regadenoson stress SPECT imaging. Imaging was conducted with one of two radiotracers (99mTc sestamibi or tetrofosmin). Regadenoson 0.4 mg was administered prior to stress SPECT as a single bolus injection.
- MDCT: Multidetector Computed Tomography (MDCT), composed of CCTA and regadenoson CTP. Regadenoson stress CTP was performed prior to rest CCTA/CTP imaging. Regadenoson 0.4 mg was administered prior to stress CTP as a single bolus injection. The rest CCTA/CTP was performed at least 30 minutes after completion of the stress CTP, after resolution of any symptoms brought on by the regadenoson infusion and after the participant's heart rate had returned to baseline.
Arm/Group | SPECT | MDCT
Serious Adverse Events (participants affected / at risk) | 1/117 | 0/116
Other Adverse Events (participants affected / at risk) | 53/117 | 59/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPECT (N=117) | MDCT (N=116)
Gastritis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPECT (N=117) | MDCT (N=116)
Headache (Nervous system disorders) | 15 | 23
Dizziness (Nervous system disorders) | 11 | 6
Flushing (Vascular disorders) | 18 | 26
Nausea (Gastrointestinal disorders) | 9 | 6
Angina pectoris (Cardiac disorders) | 4 | 9
Chest discomfort (General disorders) | 11 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 10

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.